CLINICAL TRIAL: NCT02873169
Title: Interest of Implantable Cardioverter-defibrillator in Primary Prevention in Patient With Continuous Flow Left Ventricular Assist Device (CF-LVAD)
Brief Title: Determination of Risk Factors of Ventricular Arrhythmias (VAs) After Implantation of Continuous Flow Left Ventricular Assist Device With Continuous Flow Left Ventricular Assist Device (CF-LVAD)
Acronym: ASSIST-ICD
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC15_8806_ASSIST-ICD
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-02

CONDITIONS: Severe Cardiac Insufficiency
Keywords: Left ventricular assist device; Ventricular Arrhythmias; Implantable Cardioverter-defibrillator
MeSH Terms: conditions — Heart Failure | interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Implantable cardioverter-defibrillator — Collection of clinical, biological, hemodynamic and rhythmic data

SUMMARY:
Determination of risk factors of ventricular arrhythmias (VAs) after implantation of continuous flow left ventricular assist device in order to characterize which patient requires ICD implantation in primary prevention.

ELIGIBILITY:
Inclusion Criteria:

* Patient above 18 years old
* Patients with CF-LVAD with or without ICD

Exclusion Criteria:

* Patients subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with continuous flow left ventricular assist device
Sampling Method: Probability Sample
Enrollment: 681 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of early VAs (<30 days post operatively) and late VAs (>30 days post operatively) in patient with CF-LVAD with or without ICD | 30 days
  Clinical, biological, hemodynamic and rhythmic data

SECONDARY OUTCOMES:
Mortality in patients with CF-LVAD with or without VAs | 30 days
Mortality in patients with CF-LVAD with or without ICD | 30 days

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - CHU de Bordeaux, Bordeaux
  - Hospices Civils de Lyon - Hôpital Louis Pradel, Bron
  - CHU de Caen, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - Centre chirurgical Marie-Lannelongue, Le Plessis-Robinson
  - CHRU de Lille, Lille
  - AP-HM - Hôpital de la Timone, Marseille
  - CHRU de Montpellier, Montpellier
  - CHRU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - Hôpital Européen Georges Pompidou, Paris
  - APHP - Hôpital Bichat, Paris
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Charton M, Flecher E, Leclercq C, Delmas C, Dambrin C, Goeminne C, Vincentelli A, Michel M, Lehelias L, Verdonk C, Para M, Pozzi M, Obadia JF, Boignard A, Chavanon O, Barandon L, Nubret K, Kindo M, Minh TH, Gaudard P, Pelce E, Gariboldi V, Litzler PY, Anselme F, Babatasi G, Belin A, Garnier F, Bielefeld M, Hamon D, Lellouche N, Bourguignon T, Genet T, Eschalier R, D'Ostrevy N, Bories MC, Jouan J, Vanhuyse F, Blangy H, Doucerain J, Martins RP, Galand V. Suicide Attempts Among LVAD Recipients: Real-Life Data From the ASSIST-ICD Study. Circulation. 2020 Mar 17;141(11):934-936. doi: 10.1161/CIRCULATIONAHA.119.041910. Epub 2020 Mar 10. No abstract available. PMID 32153210
- [Derived] Galand V, Flecher E, Auffret V, Pichard C, Boule S, Vincentelli A, Rollin A, Mondoly P, Barandon L, Pernot M, Kindo M, Cardi T, Gaudard P, Rouviere P, Senage T, Jacob N, Defaye P, Chavanon O, Verdonk C, Ghodbane W, Pelce E, Gariboldi V, Pozzi M, Obadia JF, Savoure A, Anselme F, Babatasi G, Belin A, Garnier F, Bielefeld M, Hamon D, Lellouche N, Pierre B, Bourguignon T, Eschalier R, D'Ostrevy N, Bories MC, Marijon E, Vanhuyse F, Blangy H, Verhoye JP, Leclercq C, Martins RP. Early Ventricular Arrhythmias After LVAD Implantation Is the Strongest Predictor of 30-Day Post-Operative Mortality. JACC Clin Electrophysiol. 2019 Aug;5(8):944-954. doi: 10.1016/j.jacep.2019.05.025. Epub 2019 Aug 19. PMID 31439296
- [Derived] Martins RP, Leclercq C, Bourenane H, Auffret V, Boule S, Loobuyck V, Dambrin C, Mondoly P, Sacher F, Bordachar P, Kindo M, Cardi T, Gaudard P, Rouviere P, Michel M, Gourraud JB, Defaye P, Chavanon O, Kerneis C, Ghodhbane W, Pelce E, Gariboldi V, Pozzi M, Grinberg D, Litzler PY, Anselme F, Babatasi G, Belin A, Garnier F, Bielefeld M, Hamon D, Lellouche N, Pierre B, Bourguignon T, Eschallier R, D'Ostrevy N, Bories MC, Jouan J, Vanhuyse F, Sadoul N, Flecher E, Galand V. Incidence, predictors, and clinical impact of electrical storm in patients with left ventricular assist devices: New insights from the ASSIST-ICD study. Heart Rhythm. 2019 Oct;16(10):1506-1512. doi: 10.1016/j.hrthm.2019.06.021. Epub 2019 Jun 27. PMID 31255846
- [Derived] Tattevin P, Flecher E, Auffret V, Leclercq C, Boule S, Vincentelli A, Dambrin C, Delmas C, Barandon L, Veniard V, Kindo M, Cardi T, Gaudard P, Rouviere P, Senage T, Jacob N, Defaye P, Chavanon O, Verdonk C, Para M, Pelce E, Gariboldi V, Pozzi M, Grinberg D, Savoure A, Litzler PY, Babatasi G, Belin A, Garnier F, Bielefeld M, Hamon D, Lellouche N, Bernard L, Bourguignon T, Eschalier R, D'Ostrevy N, Jouan J, Varlet E, Vanhuyse F, Blangy H, Martins RP, Galand V. Risk factors and prognostic impact of left ventricular assist device-associated infections. Am Heart J. 2019 Aug;214:69-76. doi: 10.1016/j.ahj.2019.04.021. Epub 2019 May 6. PMID 31174053
- [Derived] Galand V, Flecher E, Auffret V, Boule S, Vincentelli A, Dambrin C, Mondoly P, Sacher F, Nubret K, Kindo M, Cardi T, Gaudard P, Rouviere P, Michel M, Gourraud JB, Defaye P, Chavanon O, Verdonk C, Ghodbane W, Pelce E, Gariboldi V, Pozzi M, Obadia JF, Litzler PY, Anselme F, Babatasi G, Belin A, Garnier F, Bielefeld M, Hamon D, Radu C, Pierre B, Bourguignon T, Eschalier R, D'Ostrevy N, Bories MC, Marijon E, Vanhuyse F, Blangy H, Verhoye JP, Leclercq C, Martins RP; ASSIST-ICD Investigators. Predictors and Clinical Impact of Late Ventricular Arrhythmias in Patients With Continuous-Flow Left Ventricular Assist Devices. JACC Clin Electrophysiol. 2018 Sep;4(9):1166-1175. doi: 10.1016/j.jacep.2018.05.006. Epub 2018 Jul 25. PMID 30236390